CLINICAL TRIAL: NCT03982160
Title: Role of Decreased Nitric Oxide in the Tonic Elevation of Resting Sympathetic Nerve Activity in Chronic Kidney Disease Patients
Brief Title: L-arginine to Reduce Sympathetic Nerve Activity in CKD Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas at Arlington (Other)
Responsible Party: Principal Investigator, Paul Fadel, Professor, The University of Texas at Arlington
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CKD-IRB-2016-0069
Record Dates: First submitted 2019-06-06; First posted 2019-06-11 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Chronic Kidney Disease
Keywords: L-arginine; blood pressure; ADMA
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Arginine

STUDY DESIGN:
Intervention Model Description: This will be a randomize, saline-controlled crossover design study
Who Masked: Participant
Masking Description: Subjects will receive systemic intravenous infusion of L-arginine or saline for 30 minutes in a randomized order. The randomization will be carried out by research personnel.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- L-arginine (Experimental): Intravenous infusion of L-arginine (250-350 mg/kg) will be performed for 30 minutes.
  Interventions: Drug: L-Arginine
- Saline (Placebo Comparator): Saline will be infused for 30 minutes
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: L-Arginine — Arginine Hydrochloride 60% concentration injection 15 g in 25 mL, contains arginine hydrochloride 600 mg/mL in water for injections to 25 mL.
  Arms: L-arginine
Other: Placebo — Saline
  Arms: Saline

SUMMARY:
Chronic kidney disease (CKD) is associated with a higher risk of cardiovascular disease and death. An overactive sympathetic nervous system in CKD patients is one of the major mechanisms increasing the cardiovascular risks in this patient population. A potential signal driving sympathetic nerve activity (SNA) involves accumulation of the endogenous nitric oxide synthase (NOS) inhibitor asymmetric dimethylarginine (ADMA). ADMA is elevated in CKD and is a strong, independent predictor of future cardiovascular events in these patients. .

The goal of this study is to determine whether overcoming the accumulation of endogenous ADMA with acute L-arginine infusion reduces SNA in CKD patients.

DETAILED DESCRIPTION:
The central hypothesis is that accumulation of ADMA constitutes a major mechanism for the sympathetic overactivity and hypertension in patients with CKD. In this study, the investigators will determine if restoration of NO production with the infusion of L-arginine reduces SNA and blood pressure. On the experimental day, CKD patients will arrive at the laboratory fasted with no morning meds, will refrain from caffeine for 12 hours, and alcohol and physical activity for 24 hours. The collaborating physician Dr. Ashfaq Siddiqui will review subject medications and advise regarding any withholding of medications. If Dr. Siddiqui deems that a medication should not be withheld the investigators will proceed with the patient taking the medication. Prior to any screening/testing, all experimental measurements and procedures will be explained in detail and subjects will provide written, informed consent. A medical health history questionnaire will be filled out. Women of child-bearing age will provide a urine sample for a pregnancy testing prior to any study procedures. The research nurse will place an intravenous catheter in antecubital or hand vein. Subjects will be familiarized with the experimental measures and procedures prior to actual testing. Following this, the subjects will be instrumented with ECG leads, an arterial blood pressure (BP) finger-cuff (Finometer), an arterial BP upper-arm cuff for intermittent absolute BP values, and a strain gauge pneumobelt placed around the abdomen to monitor respiratory excursions. After measuring blood pressure and pulse wave velocity using applanation tonometry, a Doppler ultrasound probe will then be positioned for beat-to-beat measurements of blood velocity and artery diameter and flow-mediated dilation (FMD) will be performed. After this, continuous recording of muscle sympathetic nerve activity (MSNA) will be obtained from the peroneal nerve of the leg, as described below. Following all instrumentation, 25 minutes of resting baseline data (continuous heart rate, MSNA, BP, respiration, and blood flow) will be collected. A blood sample will then be obtained from the intravenous catheter. Next, systemic intravenous infusion of L-arginine, at a dose of 250-350 mg/kg, or saline will be performed for 30 minutes in a randomized order. During each infusion, cardiovascular measurements (heart rate, BP and MSNA) will be recorded continuously and an FMD and cold pressor test performed. The blood draw will be repeated after L-arginine infusion. A 15-minute recovery period will be provided between infusions. Thus, for this study, patients will visit the lab once and the visit will take approximately 5 hours.

ELIGIBILITY:
Inclusion Criteria:

* CKD patients classified as Stage 3 and 4 of National Kidney Foundation Classification with estimated glomerular filtration rate (GFR) between 15 and 59 mL/min/1.73 m2 according to the Modification of Diet in Renal Disease (MDRD) formula based on serum creatinine, age, gender, and race.
* Men and women 35 to 75 years of age

Exclusion Criteria:

* myocardial infarction
* heart failure
* anemia (hemoglobin <8 g/dl)
* cancer with current treatment
* previous organ transplantation
* immunosuppressant therapy
* human immunodeficiency virus infection
* pregnancy and/or lactating
* current tobacco use
* taking menopausal drugs (estradiol)
* treatment for diabetic neuropathy
* resting heart rate ≥ 100 bpm and
* systolic blood pressure ≤ 90 mmHg

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Muscle sympathetic nerve activity (MSNA) will be reduced after L-arginine infusion | 30 minutes
  Multiunit postganglionic MSNA will be recorded using standard microneurographic techniques. Briefly, a unipolar tungsten microelectrode will be inserted into muscle fascicles of the peroneal nerve near the fibular head of the right leg. Neural signals will be amplified, filtered (bandwidth, 700-2,000 Hz), rectified, and integrated (time constant, 0.1 s) to obtain mean voltage neurograms (University of Iowa Bioengineering, Iowa City, IA).

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Fadel, PhD, Principal Investigator — University of Texas at Arlington
Locations (2):
- United States (2):
  - University of Delaware, Newark, Delaware
  - UT Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No